CLINICAL TRIAL: NCT00162318
Title: A Phase I Study of Cetuximab in Combination With Gefitinib in Patients With Advanced/Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-064
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Gefitinib

ARMS (1):
- A (Experimental)
  Interventions: Drug: Cetuximab + Gefitinib

INTERVENTIONS:
Drug: Cetuximab + Gefitinib — IV solution + tablet, IV + oral, ERB (100 mg/m2, 200 mg/m2 + 250 mg/m2 IV) +GEF 250 mg tablet, ERB weekly/ GEF once daily, Until disease progression.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to find a safe and effective dose of Erbitux and Iressa for subject with non small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced or metastatic non small cell lung cancer.
* Subjects should have had at least one prior chemotherapy with a platinum based therapy.

Exclusion Criteria:

* Subjects are excluded from this study if they do not have non small cell lung cancer that is advanced or metastatic or have not had at least one prior platinum based chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Safe and effective dose of combination of Erbitux and Iressa therapy.

SECONDARY OUTCOMES:
Response will be measured by radiographic measurement of disease every 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Local Institution, Pittsburgh, Pennsylvania, United States